CLINICAL TRIAL: NCT02411851
Title: An Investigator-Initiated Study to Assess the Efficacy and Degree of Irritation of Ingenol Mebutate 0.015% Gel and Dermasil Lotion Versus Ingenol Mebuate 0.015% Alone in the Treatment of Actinic Keratoses (AK) on the Face.
Brief Title: Treatment of Actinic Keratoses (AK) on the Face
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Mark Lebwohl, Professor and System Chair Dermatology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 14-1319
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ingenol mebutate alone (Active Comparator): At Visit 1, ingenol mebutate 0.015% alone on the second 25 cm2 treatment area. The treatment area receiving ingenol mebutate 0.015% alone will apply the medication as directed per approved drug labeling. Patients will apply ingenol mebutate gel on Day 2 and Day 3.
  Interventions: Drug: ingenol mebutate 0.015%
- Ingenol mebutate and dermasil lotion (Experimental): At Visit 1, ingenol mebutate 0.015% and dermasil lotion on one 25 cm2 treatment area. The treatment area receiving both ingenol mebutate 0.015% and dermasil lotion, will first apply ingenol mebutate 0.015% allow the gel to dry completely as per drug labeling on Day 1. The patient will allow at least 6 hours between the application of ingenol mebutate and dermasil lotion on Day 2 and 3. Patients will apply dermasil lotion daily on Day 2 until at least Day 8. At Day 8, the physician will reassess whether dermasil application should be continued to Day 15 or ceased. At Day 15, the physician will reassess whether dermasil application should be continued to Day 29 or ceased.
  Interventions: Drug: ingenol mebutate 0.015%; Other: dermasil lotion

INTERVENTIONS:
Drug: ingenol mebutate 0.015% — one cycle of ingenol mebutate 0.015% on two 25 cm2 treatment areas
Other: dermasil lotion — Dermasil lotion has 1% dimethicone as its active ingredient - part of the family of silicone oils, is a hypoallergenic, noncomedogenic, and nonacnegenic agent
  Arms: Ingenol mebutate and dermasil lotion

SUMMARY:
Actinic keratoses (AK) are common cutaneous lesions associate with chronic ultraviolet radiation exposure. While most authorities consider AK as a pre-malignant lesion, some consider it as an incipient squamous cell carcinoma (SCC). Ingenol mebutate is the active compound in the sap from Euphorbia peplus L. (E. peplus). Topical ingenol mebutate treatment has been approved for the treatment of AKs. Ingenol mebutate gel 0.015% has shown to not only have a high clearance rate but also a transient localized inflammatory skin response that resolves quickly without sequelae. However, these localized skin responses (eg erythema, erosion/ulceration, edema, etc.) can often be unpleasant and unsightly. Currently, there are no clinical studies evaluating combination therapies (eg topical steroids, emollients) with ingenol mebutate 0.015% that would decrease irritation and improve wound healing while maintaining efficacy.

DETAILED DESCRIPTION:
Actinic keratoses (AK) are common cutaneous lesions associate with chronic ultraviolet radiation exposure. Ultraviolet radiation produces local and systemic immunosuppression, mutations in the p53 tumor suppressor gene, and deoxyribonucleic acid pyrimidine covalent dimmers, each of which is believed to contribute to the dysplasia seen in AK. While most authorities consider AK as a pre-malignant lesion, some consider it as an incipient squamous cell carcinoma (SCC). The risk for progression to SCC for an individual AK is reportedly low but highly variable; however, as patients often have multiple AKs, the overall risk for progression over a lifetime can be significant; thus treatment of AKs is warranted. In addition, the skin around clinically obvious AK lesions has been subject to the same chronic ultraviolet exposure, resulting in genetic damage and mutations, resulting in "field cancerization." Subclinical AKs may progress to clinical AKs, or even de novo invasive SCCs.

Among the current therapies for the treatment of AK are excisional surgery, cryosurgery, electrodesiccation and curettage, topical chemotherapy and light therapies. Cryosurgery is considered the gold standard for therapy, however as with other lesion-directed therapies, cryosurgery does not treat subclinical lesions in the surrounding skin. Treated lesion clearance rates at 3 months post-treatment after double-freeze thaw cryotherapy has been reported to be around 76-88%; however, new lesions in the treatment field were not included. Overall lesion clearance rate, including new subclinical lesions, at approximately 5 months post-cryosurgery has been reported to be 35-51%. The inability to treat subclinical lesions with lesion-directed cryosurgery, has spurred the emergence of topical medications such as ingenol mebutate for field-directed therapy.

Ingenol mebutate is the active compound in the sap from Euphorbia peplus L. (E. peplus). The sap from E. peplus has a long history of community use for the topical treatment of various skin conditions, including AKs. Ingenol mebutate, in a gel formulation referred to as PEP005 (ingenol mebutate) Gel or PEP005 Gel, has been evaluated in clinical trials as field therapy for the topical treatment of AK and photo damaged skin and as lesion-specific treatment for seborrheic keratosis and non-melanoma skin cancer (NMSC). The mechanism of action of ingenol mebutate in AK therapy is not yet fully understood. In vivo and in vitro models have demonstrated both an induction of local lesion cell death and promotion of lesion-specific inflammatory response. A 0.015% topical formulation has been approved for the treatment of AKs in the US as a once a day for three consecutive days regimen. Topical ingenol mebutate treatment may also reduce subclinical lesions in the treatment area, resulting in fewer "new" AK lesions developing over the same period of time when compared to focal treatment.

Phase III data demonstrated complete field clearance of AKs in 37-47% on the face as well as sustained clearance of approximately 50% twelve months post treatment. Similarly a randomized controlled study found a mean reduction of 83% in AK lesions on the face. 87.2% of AK's in the treatment area at baseline were still clear 12 months later. Previous clinical studies report mild to moderate local adverse events (AE) such as pruritus, pain, irritation and local skin response (LSR) (eg erythema, flaking, scaling). The unpleasant and often unsightly localized skin irritation can be emotionally difficulty for patients and provoke anxiety. It is unknown whether a large inflammatory reaction is necessary for successful treatment of actinic keratosis with ingenol mebutate 0.015%. Currently, there are no clinical studies evaluating combination therapies (eg topical steroids, barrier creams, etc.) with ingenol mebutate 0.015% that would decrease irritation while maintaining efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old.
* Subjects must be in good general health as confirmed by the medical history.
* Subjects must be able to read, sign, and understand the informed consent
* Subjects must have two separate, relatively symmetrical 25 cm2 treatment areas on the face with at least 3-8 non-hypertrophic AKs.
* Subject must be willing to forego any other treatments on the face, including tanning bed use and excessive sun exposure while in the study.
* Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods and to comply with all study requirements including concomitant medication and other treatment restrictions.
* If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

* Subjects with a history of melanoma anywhere on the body.
* Subjects with an unstable medical condition as deemed by the clinical investigator.
* Subjects with current non-melanoma skin cancer on the face.
* Subjects with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of AKs.
* Subjects who have previously been treated with ingenol mebutate: on the face in the past 6 months; or outside of the study area within the past 30 days.
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc).
* Subjects who have active chemical dependency or alcoholism as assessed by the investigator.
* Subjects who have known allergies to any excipient in the ingenol mebutate 0.015% gel and/or dermasil lotion.
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device on the study area within 30 days prior to study treatment initiation.
* Subjects who have received any of the following within 90 days prior to study treatment initiation:

  * interferon or interferon inducers
  * cytotoxic drugs
  * immunomodulators or immunosuppressive therapies (inhaled/ intranasal steroids are permitted)
  * oral or parenteral corticosteroids
  * topical corticosteroids if greater than 2 gm/day
  * any dermatologic procedures or surgeries on the study area (including any AK treatments)
* Subjects who have used any topical prescription medications on the study area within 30 days prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Local Skin Reaction (LSR) | up to day 57
  Investigator assessment of the degree of irritation as measured by local skin reactions at day 57 as compared to baseline.

SECONDARY OUTCOMES:
AK lesion count | baseline and day 57
  Change in the number of AK lesions at 57 days as compared to baseline to assess AK clearance
Visual Analog Scale (VAS) Survey | baseline and day 57
  The patient pruritus VAS survey to assess patient treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States